CLINICAL TRIAL: NCT07128407
Title: The Effect of Radiation Protection Training Based on Protection Motivation Theory on Nurses' Knowledge, Awareness, Motivation and Safety Behaviors: A Randomized Controlled Trial.
Brief Title: PMT-Based Radiation Safety Training for Nurses: Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Mahmut AY, PhD Student, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NEU-MAY-2025-01
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Occupational Radiation Exposure in Operating Room Nurses
Keywords: Radiation Protection; Occupational Safety; Nursing Safety Behavior; Occupational Radiation Exposure; Protection Motivation Theory; Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: he study involves 54 operating room nurses randomly assigned to either the experimental group (n=27) receiving a Protection Motivation Theory-based radiation protection training, or the control group (n=27) not receiving the intervention during the study period. Outcomes including knowledge, awareness, motivation, and safety behaviors are assessed before and after the intervention to evaluate the effectiveness of the training program.
Masking Description: No masking is applied in this study; both participants and investigators are aware of group assignments (open label).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants receive a structured radiation protection training program based on Protection Motivation Theory (PMT). The program targets threat appraisal (perceived severity and vulnerability) and coping appraisal (response efficacy, self-efficacy, and response cost) processes to improve nurses' knowledge, awareness, motivation, and safety behaviors. Outcomes are assessed before and after the intervention.
  Interventions: Behavioral: Protection Motivation Theory-Based Radiation Protection Training
- Control Group (No Intervention): Participants do not receive any intervention during the study period. They continue their routine clinical practice. Outcomes are assessed at the same time points as the experimental group to allow comparison.

INTERVENTIONS:
Behavioral: Protection Motivation Theory-Based Radiation Protection Training — A structured educational program designed according to Protection Motivation Theory (PMT). The program targets both threat appraisal (perceived severity and vulnerability) and coping appraisal (response efficacy, self-efficacy, and response cost) processes to improve nurses' knowledge, awareness, motivation, and safety behaviors regarding radiation protection.
  Arms: Experimental Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a Protection Motivation Theory (PMT)-based radiation protection training program on nurses' knowledge, awareness, motivation, and safety behaviors. The study includes 54 operating room nurses randomly assigned to experimental (n=27) and control (n=27) groups. The intervention targets both threat appraisal (perceived severity and vulnerability) and coping appraisal (response efficacy, self-efficacy, and response cost) processes. It is hypothesized that PMT-based training will improve nurses' radiation protection knowledge, increase awareness, strengthen motivation, and enhance safety behaviors. The findings are expected to contribute to nursing curricula, institutional radiation safety policies, and the development of a safety culture in healthcare settings.

DETAILED DESCRIPTION:
The increasing use of ionizing radiation in medical procedures has raised concerns about occupational exposure among healthcare professionals, including nurses, who may be directly or indirectly exposed during their clinical duties. Evidence from the literature indicates that nurses often have insufficient knowledge and awareness regarding radiation protection, which may lead to suboptimal safety practices and increased health risks. Enhancing radiation safety among nurses is crucial for both occupational health and patient safety.

Protection Motivation Theory (PMT), developed by Rogers, provides a comprehensive framework for understanding and influencing health-related protective behaviors. PMT posits that behavior change is influenced by two cognitive processes: threat appraisal (perceived severity and perceived vulnerability) and coping appraisal (response efficacy, self-efficacy, and response cost). Educational interventions structured according to PMT can effectively promote protective health behaviors by addressing both risk perception and the perceived ability to perform protective actions.

This randomized controlled trial aims to evaluate the effectiveness of a PMT-based radiation protection training program in improving nurses' knowledge, awareness, motivation, and safety behaviors related to radiation protection. A total of 54 operating room nurses will be randomly assigned to either the experimental group (n=27), which will receive structured PMT-based radiation safety education, or the control group (n=27), which will not receive the intervention during the study period. The training program targets both threat and coping appraisal processes and is delivered in a structured format designed to address the cognitive and behavioral components of radiation safety.

Primary and secondary outcome measures will be assessed before and after the intervention using validated instruments. The primary outcome is the change in radiation protection behavior scores, while secondary outcomes include changes in knowledge, awareness, and motivation scores. It is hypothesized that the intervention group will demonstrate significant improvements in all outcome measures compared to the control group.

The results of this study are expected to inform the integration of radiation safety content into nursing curricula, guide the development of institutional policies on radiation protection, and contribute to fostering a culture of safety in healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses working in the operating room or intervention areas where ionizing radiation is used.
* Willing to participate and provide informed consent.
* Able to attend the full radiation protection training program (for the experimental group).

Exclusion Criteria:

* Nurses not working in areas with exposure to ionizing radiation.
* Nurses who have previously received formal radiation protection training within the last 12 months.
* Inability to complete the study questionnaires or training program due to language or cognitive barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-07 (Estimated); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Change in Radiation Protection Knowledge | Pre-intervention, Immediate Post-intervention, and 1 Month Post-intervention
  Assessed using a validated Radiation Protection Knowledge Questionnaire specifically developed for nurses. The measure evaluates participants' understanding of radiation risks, protection methods, and safe practices.

SECONDARY OUTCOMES:
Change in Radiation Protection Awareness | Pre-intervention, Immediate Post-intervention, and 1 Month Post-intervention
  Evaluated with a standardized awareness scale assessing nurses' perception of radiation hazards and the need for protection
Change in Protection Motivation | Pre-intervention, Immediate Post-intervention, and 1 Month Post-intervention
  Measured using a Protection Motivation Theory-based scale capturing threat appraisal and coping appraisal dimensions.
Change in Safety Behaviors | Pre-intervention, Immediate Post-intervention, and 1 Month Post-intervention
  Assessed via a self-reported Radiation Protection Behavior Scale, evaluating adherence to safety protocols in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: BİLGEN ÖZLÜK, Assoc. Prof. Dr., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University Faculty of Medicine Hospital, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No